CLINICAL TRIAL: NCT05335044
Title: An Open-label, Randomized, Single-dose, 2-sequence, 4-period, Cross-over, Phase 1 Study to Evaluate the Safety and Pharmacokinetics of CKD-331 in Healthy Adult Volunteers
Brief Title: Study to Evaluate the Safety and Pharmacokinetics of CKD-331
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: A124_01BE2203
Record Dates: First submitted 2022-04-12; First posted 2022-04-19 (Actual); Last update posted 2023-06-09 (Actual); Status verified 2023-06

CONDITIONS: Hypertension and Dyslipidemia
MeSH Terms: conditions — Hypertension; Dyslipidemias

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sequence A (Experimental): Period 1: EX5619 - A single oral dose of 1 tablet under fasting condition
  Period 2: CKD-331 - A single oral dose of 2 tablets under fasting condition
  Period 3: EX5619 - A single oral dose of 1 tablet under fasting condition
  Period 4: CKD-331 - A single oral dose of 2 tablets under fasting condition
  Interventions: Drug: CKD-331; Drug: EX5619
- Sequence B (Experimental): Period 1: CKD-331 - A single oral dose of 2 tablets under fasting condition
  Period 2: EX5619 - A single oral dose of 1 tablet under fasting condition
  Period 3: CKD-331 - A single oral dose of 2 tablets under fasting condition
  Period 4: EX5619 - A single oral dose of 1 tablet under fasting condition
  Interventions: Drug: CKD-331; Drug: EX5619

INTERVENTIONS:
Drug: CKD-331 — QD, PO
Drug: EX5619 — QD, PO

SUMMARY:
Phase 1 study to evaluate the safety and pharmacokinetics of CKD-331 in healthy adult volunteers

DETAILED DESCRIPTION:
An open-label, randomized, single-dose, 2-sequence, 4-period, cross-over, phase 1 study to evaluate the safety and pharmacokinetics of CKD-331 in healthy adult volunteers

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult volunteers aged ≥ 19 years
2. Weight ≥55kg with calculated body mass index (BMI) of 18 to 30 kg/m2
3. Those who have no congenital diseases or chronic diseases and have no abnormal symptoms or findings.
4. Those who are eligible for clinical trials based on laboratory (hematology, blood chemistry, serology, urology) and 12-lead ECG results at screening.
5. Those who agree to contraception during the participation of clinical trial.
6. Individuals who voluntarily decide to participate and agree to comply with the cautions after fully understand the detailed description of this clinical trial.

Exclusion Criteria:

1. Those who have no medical history of digestive disease, cardiovascular disease, endocrine disease, respiratory system, blood·tumor disease, infection disease, nephrology disease, genitourinary disease, neuron disease, skeletal disease, immunological disease, otolaryngological disease, dermatological disease, ophiological disease
2. Those who have a history of gastrointestinal surgery except simple appendectomy and hernia surgery.
3. Those who take barbiturate and any related drugs which may cause induction or inhibition of drug metabolism within 1 month before the first administration of investigational products.
4. Those who received investigational products or participated in bioequivalence tests within 6 months before the first administration of clinical trial drugs.
5. Those who donated whole blood or apheresis within 8 weeks or 4 weeks respectfully, or received blood transfusion within a month.
6. Those who exceed an alcohol and cigarette consumption than below criteria Alcohol

   * Man: 21 glasses/week
   * Woman: 14 glasses/week (1 glass: Soju 50mL, Wine 30mL, or beer 250mL) Smoking: 20 cigarettes/day
7. Those who have genetic problems such as galactose intolerance, Lapp lactose deficiency or glucose-galactose malabsorption.
8. Those who are deemed insufficient to participate in this clinical study by investigators.
9. Woman who are pregnant or breastfeeding.

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2022-05-31 (Actual); Primary Completion 2022-06-23 (Actual); Study Completion 2022-07-12 (Actual)

PRIMARY OUTCOMES:
Cmax of CKD-331 | Pre-dose (0 hour), 0.17, 0.33, 0.5, 0.67, 0.83, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 34 hours
  Cmax: Maximum plasma concentration of the drug
AUCt of CKD-331 | Pre-dose (0 hour), 0.17, 0.33, 0.5, 0.67, 0.83, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 34 hours
  AUCt: Area under the concentration-time curve from time zero to time

CONTACTS AND LOCATIONS:
Overall Officials: Jaewoo Kim, M.D., PhD., Principal Investigator — Yanhji Hospital
Locations (1):
- H plus Yangji hospital, Seoul, South Korea